CLINICAL TRIAL: NCT03868293
Title: Low Intensity Focused Ultrasound Treatment for Epilepsy: A Pilot Trial
Brief Title: Low Intensity Focused Ultrasound Epilepsy: A Pilot Trial
Acronym: LIFUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ellen J Bubrick, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018P000125
Record Dates: First submitted 2019-02-08; First posted 2019-03-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Drug-Resistant Epilepsy (temporal lobe) (Experimental): Pulsed low intensity focused ultrasound
  Interventions: Device: Focused ultrasound

INTERVENTIONS:
Device: Focused ultrasound — Pulsed low intensity focused ultrasound

SUMMARY:
The aim of the proposed pilot study is to investigate patient tolerability and efficacy of moderate term, repeated exposure of Pulsed Low-Intensity Focused Ultrasound (PLIFUS) in patients with drug-resistant temporal lobe epilepsy.

DETAILED DESCRIPTION:
The aim of the proposed pilot study is to investigate safety and tolerability of moderate term, repeated exposure of Pulsed Low-Intensity Focused Ultrasound (PLIFUS) in patients with drug-resistant temporal lobe epilepsy.

Due to the lack of options for patients with drug-resistant epilepsy, investigations into alternative noninvasive treatments are warranted. PLIFUS has been shown to safely modulate neuronal tissue, and is non-invasive and painless. Several human studies have shown that the use of PLIFUS can suppress somatosensory evoked potentials and induce functional magnetic resonance imaging (MRI) responses.

Once the subject is enrolled in the study, the subject will be scheduled for a standard brain MRI scan at BWH if they have not had one in the last 3 months. The subject will be asked to keep track of their seizure events in the Daily Seizure Log Diary from the screening visit until 6 months after the last treatment session.

The treatment period will include 6 treatment sessions total. These will occur 2 days per week for 3 weeks, each lasting approximately 1-2 hours, starting 1 month after seizure logging begins.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least eighteen (18) years of age
* Subjects with drug-resistant temporal lobe epilepsy whose seizures involve altered awareness (ie failed at least two trials of antiepileptic drugs for seizures), as determined by one of the BWH epilepsy neurologists based on clinical seizure semiology and/or EEG findings.
* Subjects who experience at least 1-2 seizures per month on average, are aware of or have reliable caregivers who are aware of when seizures occur and can reliably log seizure frequency
* Subjects who have the cognitive ability to read and understand the consent form, describe any potential symptoms experienced during or after treatments.

Exclusion Criteria:

* Subjects with a cognitive or psychiatric disorder that limits the ability to give informed consent or are unable to cooperate with testing
* Subjects with dementia or other progressive degenerative disease, delirium or active psychosis
* Subjects with ferromagnetic materials in the head
* Subjects with severe cardiac disease, increased intracranial pressure, or a Transcutaneous Electrical Nerve Stimulation (TENS) unit
* Subjects who have primary generalized epilepsy or non-epileptic seizures
* Subjects who have experienced status epilepticus in the 3 months leading up to enrollment in the study
* Subjects (females) who are pregnant, or are of childbearing potential and not willing to use reliable birth control during the treatment period.
* Subjects who are unable to get a brain MRI for any reason (implanted metal in body, inability to lie still)
* Subjects with current brain tumors or an intracranial vascular lesion
* Subjects with severe, uncontrolled medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation.
* Subjects with holes in the treatment area of the skull from trauma or prior surgery
* Subjects with pacemakers, medication pumps, and other implanted electronic hardware. If a subject has a working Vagal Nerve Stimulator in place, the device will be turned off prior to each treatment session and then turned back on after each session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Patient tolerability of moderate term, repeated exposure toPulsed Low-Intensity Focused Ultrasound (PLIFUS) (Adverse Events assessment) | 3 months
  The aim of the proposed pilot study is to investigate patient tolerability of moderate term, repeated exposure of Pulsed Low-Intensity Focused Ultrasound (PLIFUS) in patients with drug-resistant temporal lobe epilepsy. We hypothesize that the treatments will be well-tolerated, without adverse events.
Efficacy of PLIFUS in reducing seizure frequency | 3 months
  The aim of the proposed pilot study is to investigate patient efficacy of moderate term, repeated exposure of Pulsed Low-Intensity Focused Ultrasound (PLIFUS) in patients with drug-resistant temporal lobe epilepsy .We hypothesize that PLIFUS stimulation will result in mechanical disruption of the target tissue (here, the epileptogenic focus), preserving the integrity of the tissue but rendering it unable (or less able) to mount seizure activity for a period of time.
  We, therefore, will assess improvement in subjects' seizure frequency by evaluating seizure frequency during and 30 days after the treatment period relative to a 30 day pre-treatment baseline period.
Effect of PLIFUS on patient EEG (evaluate number of attenuated epileptiform discharges) | 3 months
  We hypothesize that subjects' EEGs will show improvement (fewer and/or attenuated epileptiform discharges). Study Epileptologists (either the PI or Co-I) will interpret EEG results during the first and last treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen J Bubrick, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bubrick EJ, McDannold NJ, White PJ. Low Intensity Focused Ultrasound for Epilepsy- A New Approach to Neuromodulation. Epilepsy Curr. 2022 Mar 29;22(3):156-160. doi: 10.1177/15357597221086111. eCollection 2022 Jun. PMID 36474831

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT03868293/Prot_SAP_000.pdf